CLINICAL TRIAL: NCT05624541
Title: Investigation of the Turkish Validity and Reliability of Specific Test of Early Infant Motor Performance (STEP) in Follow-Up of Risk Infants
Brief Title: Validity and Reliability of Specific Test of Early Infant Motor Performance (STEP) Version 3.0
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2021.887
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-10

CONDITIONS: Preterm Birth Complication; Cerebral Palsy; Infant, Premature, Diseases
Keywords: infant; validity and reliability; premature
MeSH Terms: conditions — Cerebral Palsy; Infant, Premature, Diseases; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- preterm Infant: 30 premature infants with a gestational age of 37 weeks and below and a history of stay in the neonatal intensive care unit will be evaluated.
  Interventions: Diagnostic Test: Measurements

INTERVENTIONS:
Diagnostic Test: Measurements — All infants at high risk of cp will be assessed by Specific Test of Early Infant Motor Performance (STEP) Version 3.0 at term age and at corrected age 3 months, by Hammersmith Infant Neurological Examination (HINE) a corrected age 3 and 6 months, also BAYLEY-III Infant and Toddler Development Assessment Scale (BAYLEY-III) at corrected 6 months.
  Other Names: Measurements of neurological development.

SUMMARY:
Cerebral palsy and other neuromotor disorders are more common in babies born preterm (<37 weeks of gestation), due to various biological and environmental risk factors and the risk increases as the gestational age decreases. Earlier and more frequent screening with the use of developmental skills tests facilitates referral to early intervention programs. Current guidelines recommend using some combination of neuroimaging and neurological examination and assessments such as neonatal imaging, general movements (GMs), and Hammersmith Infant Neurological Examination (HINE) for early diagnosis and intervention.

DETAILED DESCRIPTION:
The aim of study was to evaluate the risk of premature and low birth weight babies with the Early Infant Motor Evaluation Test (STEP), to measure the correlation of the STEP test with Bayley Infant Development Scales (Bayley-III) and Hammersmith Infant Neurological Examination (HINE) evaluations, to investigate the validity and reliability of the STEP test in the evaluation and follow-up of babies at risk.

The Early Infant Motor Evaluation Test (STEP) provides a quantitative assessment of tone and movements that allows developmental monitoring with a short screening test in terms of practical patient flow. A standardized test provides an opportunity to recognize early abnormalities in tone and movement patterns and seek treatment before milestones are delayed or abnormal movements stabilized. STEP can be used to measure early movement problems in high-risk infants, refer these infants earlier, and then monitor response to targeted interventions. It is thought that STEP can identify infants at risk of delay, thus enabling earlier initiation of targeted therapy. The implementation and scoring of STEP takes approximately 10 minutes. It does not require special training, is easy to access, is a short and fast performing neuromotor examination. As a screening test for early intervention, it can be applied in neonatal intensive care units and follow-up clinics prior to discharge, potentially improving long-term outcomes.

Technological advances in neonatal-perinatal medicine have led to a steady increase in the survival rate of preterm infants. Although the increase in survival rate has been a remarkable achievement, children born prematurely are at high risk for brain damage and long-term neurodevelopmental deficits. Premature children may have abnormal muscle tone or movements, cognitive deficits, language disorders, and behavioral problems.

Babies born preterm (<37 weeks of gestation) are three to four times more at risk for a range of motor disorders than the general population due to various biological and environmental risk factors. This highlights the need for improved surveillance and intervention strategies in this group of children.

The main goal of developmental surveillance in infants with risk factors for cerebral palsy and other neuromotor disorders is to screen for signs of delayed motor development so that physical therapy can be started as early as possible. Neuroimaging is expensive and does not detect all infants at high risk. Parental reporting of motor milestones in the first trimester is unlikely to be as accurate as methods based on direct observation. Barriers to implementing highly sensitive assessments based on direct observation include the cost of training, lack of reliability in various professions, and the duration of assessment. Most of the screening tests used involve long-term use that may harm newborns.

Accurate assessment of motor performance in infants born prematurely or with other perinatal complications requires the use of validated tests to identify delay or neurological impairment. Documenting the construct validity of a new assessment requires research that demonstrates its relevance to other tests available for similar purposes.

Recent studies also advocate the use of a combination of assessment tools in the first year of life. Studies have proven that the use of a combination of standard neurologic and motor assessments for early diagnosis and intervention in the evaluation of at-risk infants is more effective.

It is known that the STEP test does not require certification training and whose reliability is valid, does not have a Turkish version.In this thesis, the validity and reliability of the Early Infant Motor Evaluation Test (STEP) will be investigated, and its correlation with the Hammersmith Infant Neurological Examination (HINE) and Bayley Infant Development Scales (Bayley-III) evaluation will be evaluated. The translation of the scale into Turkish will be carried out separately by two health professionals who are fluent in the original language and medical terminology. The final version of the scale will be translated back from the target language to the original language by a sworn translator who has no knowledge of the subject, and the back translation will be compared with the original questionnaire.

Medical records and demographic data of the patients whose verbal and written consents were obtained will be obtained and STEP test will be applied at term age and at 3 months, with HINE test at corrected 3 months and 6 months and Bayley III test at corrected 6 month.

ELIGIBILITY:
Inclusion Criteria:

1. Babies born before <37 weeks of gestation and treated in the neonatal intensive care unit
2. Infants with neurologic abnormalities (muscle hypertonia, hypotonia, hyperarousal, and abnormal general movements or cranial ultrasound abnormalities) at moderate to high risk of cerebral palsy
3. Infants referred to physiotherapy due to motor developmental delay and neurological dysfunction
4. Babies whose age range is between 0-12 months (corrected age will be calculated for premature babies)
5. Being diagnosed as a neurologically and developmentally risky baby
6. Babies who have completed medical treatments and are not in neonatal intensive care
7. Infants of families of infants who agreed to participate in the study and approved the informed consent form

Exclusion Criteria:

1. Babies with congenital cyanotic heart problems or cystic fibrosis
2. Babies with genetic disease or congenital anomalies
3. Infants on ventilator
4. Babies of families who do not accept to work

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 30 infants will be included in the study. Based on the data of the previous study, the number of participants to be included in the study was found to be correlated with G*Power 3.1.9.2 (Correlation: Bivariate) as p H1=0.89. The minimum number of individuals to be included in the sample of this study was calculated by taking effect size=0.60, α=0.05 and power=0.95, and it was found to be 30 in total. Since the effect size obtained from the sample study is large, it was preferred to use the correlation p H1=0.6 size in order to reach a larger sample size.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-18 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Specific Test of Early Infant Motor Performance (STEP) Version 3.0 | Change from term age of infants (40 weeks) to 3 month
  The STEP test is a 10-item neurodevelopmental assessment that does not require special training, evaluating infants from term to corrected 3 months for rapid and early detection of motor problems. It evaluates the infant not only by the presence or absence of motor skills, but by the quality of movement. A term cut-off score of 16 or less and a three-month cut-off score of 22 or less are important criteria in developmental delay.
Hammersmith Infant Neurological examination (HINE) | Change from the baseline of the HINE score at corrected age 3, 6th month of infants
  It is a neurodevelopmental assessment test accessible to all clinicians used for infants 2 to 24 months old. It is a 26-item test with a maximum score of 78 scored between 0-3. It has 3 sections: (1) neurological examination (26 items, scored) evaluating cranial nerve function, posture, movements, tone, reflexes, and reactions, (2) motor milestones (8 items, unscored), and (3) behaviour (3 items, unscored). Higher score indicates good neurological function.
Bayley Scales of Infant and Toddler Development (BSID -III) | Change from the baseline of the BAYLEY-III score at corrected age 6th month of infants
  It is applied to evaluate the development in cognitive, language and movement areas in children whose corrected age is between 0-42 months. Movement scale consists of two parts as fine motor and gross motor. A score below 70 is a criterion for developmental delay.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag-Saygi, Prof, Study Director — Marmara University
Locations (1):
- Marmara University Pendik Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No